CLINICAL TRIAL: NCT06191146
Title: Factors for Impairment of Renal Graft Function in Intensive Care
Acronym: RENAGRAF
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Gibot Sébastien, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023PI048
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Graft Failure; Dialysis; Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
hypothesis = hospitalization in the intensive care unit (ICU) has an impact on the outcome of the renal graft, due to the therapeutic and exploratory procedures performed.

the aim is to identify risk factors for renal graft degradation in the ICU up to 2 years after hospitalization.

Optimization of renal graft management in the ICU and management by nephrologists after the ICU

ELIGIBILITY:
Inclusion Criteria:

* kidney graft
* > 18 years
* first hospitalization in ICU

Exclusion Criteria:

* chronic hemodialysis before ICU
* transfer to intensive care immediately after transplant within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: non-dialyzed kidney transplant patient hospitalized in intensive care unit
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
composite: return to dialysis, decline in GFR < 15 ml/min, death at 2 years | 2 years after ICU
  Death within 2 years, glomerular filtration rate < 15mL/min, need for dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GIBOT, Principal Investigator — CHU NANCY Central
Locations (1):
- CHRU Nancy, Nancy, France